CLINICAL TRIAL: NCT04217941
Title: Effect of Practical Demonstration to Use Nasal Spray and Apply Intranasal Ointment on Outcome, in Cases of Recurrent Pediatric Epistaxis
Brief Title: Effect of Practical Demonstration to Use Nasal Spray and Apply Intranasal Ointment on Epistaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Ahmed Khan, ENT consultant, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMH-06-2018
Record Dates: First submitted 2019-12-29; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Epistaxis
Keywords: Epistaxis; Randomized control trial; Health education
MeSH Terms: conditions — Epistaxis; Health Education

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education with practical demonstration (Active Comparator): Participants assigned to the intervention arm received health education with practical demonstration of nasal spray and intranasal ointment .
  Interventions: Procedure: Health education with practical demonstration of nasal ointment; Drug: Health Education and practical demonstration of Nasal spray and intranasal ointment
- Health education without practical demonstration (Placebo Comparator): Participants assigned to the control arm received only health education regarding nasal spray and intranasal ointment .
  Interventions: Procedure: Health education with practical demonstration of nasal ointment

INTERVENTIONS:
Procedure: Health education with practical demonstration of nasal ointment — Health education with practical demonstration of medicine was compared to health education without practical demonstration
  Other Names: Group A and B
Drug: Health Education and practical demonstration of Nasal spray and intranasal ointment — We compared the effect of Health education and practical demonstration for using nasal spray and apply intranasal ointment compared to health education without practical demonstration
  Other Names: Health education with practical demonstration group
  Arms: Health Education with practical demonstration

SUMMARY:
To compare the result of verbally educating the parents about method of intranasal antiseptic cream application versus practically educating and demonstrating how to apply cream intra nasally.

DETAILED DESCRIPTION:
The primary outcome variables was control of epistaxis through history and clinical examination on follow up visits

ELIGIBILITY:
Inclusion Criteria:

* The children of age less than 12 years presenting with anterior recurrent epistaxis

Exclusion Criteria:

* o Children with bleeding disorders.

  * Children with liver and renal failure/dysfunction.
  * Children using anti-coagulants.
  * Those children who have gross deviated nasal septum or nasal polys etc.
  * Cases who had history of nasal injuries secondary to trauma.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
number of epistaxis episodes | 0ne month
  Success rate was measured on number of epistaxis episodes after treatment. The primary outcome variables was control of epistaxis through history and clinical examination on follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khan, MBBS, FCPS, Principal Investigator — CMH Mardan
Locations (1):
- CMH Mradan, Mardan, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No